CLINICAL TRIAL: NCT06024525
Title: Prospective, Multi-center Non-inferiority and Randomized Controlled Clinical Study to Verify Effectiveness and Safety of Paclitaxel-Coated Coronary Balloon Catheters Swide®
Brief Title: Verify Effectiveness and Safety of Paclitaxel-Coated Coronary Balloon Catheters Swide®
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP01-048B
Record Dates: First submitted 2023-08-15; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The use of a third-party independent CEC and an independent coronary angiography core laboratory to adjudicate each primary and other endpoints helps reduce measurement bias from outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel-Coated Coronary Balloon Catheters (Experimental): receiving the treatment with Swide®DCB in small vessel cohort
  Interventions: Device: Paclitaxel-Coated Coronary Balloon Catheters
- Paclitaxel-Releasing Coronary Balloon Catheter (Active Comparator): receiving the treatment with SeQuent® please Neo in small vessel cohort
  Interventions: Device: Paclitaxel-Releasing Coronary Balloon Catheters

INTERVENTIONS:
Device: Paclitaxel-Coated Coronary Balloon Catheters — to Verify Effectiveness and Safety of Paclitaxel-Coated Coronary Balloon Catheters in SVD patients
  Arms: Paclitaxel-Coated Coronary Balloon Catheters
Device: Paclitaxel-Releasing Coronary Balloon Catheters — to Verify Effectiveness and Safety of Paclitaxel-Coated Coronary Balloon Catheters in SVD patients
  Arms: Paclitaxel-Releasing Coronary Balloon Catheter

SUMMARY:
The objective of this study is to assess the safety and efficacy of the Paclitaxel-Coated Coronary Balloon Catheters Swide® (3µg/mm2 balloon surface area) in the treatment of Chinese patients with native coronary heart disease and small vessel lesions（reference diameters from 2.0mm to 2.75 mm） in comparison with Paclitaxel-Releasing Coronary Balloon Catheter SeQuent® please Neo

DETAILED DESCRIPTION:
This study conducted a prospective, multi-center, randomized controlled, non-inferiority clinical trial to compare the safety and efficacy of the Shenqi Medical paclitaxel-coated coronary balloon catheter and the paclitaxel-eluting coronary balloon catheter (SeQuent® please Neo) in the treatment of coronary artery small vascular disease.

* A total of 236 participants are planned to be recruited, and they will be allocated into the experimental group and the control group in a 1:1 ratio.
* All participants will undergo clinical follow-up at 1 month, 6 months, 9 months, 1 year, and 2 years after receiving the drug-eluting balloon angioplasty procedure.
* Angiographic re-evaluation will be conducted for all participants at 9 months after the procedure. The primary study endpoint will be the in-segment diameter stenosis in target lesion(%) at 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Related to the patients:

1. Age ≥18 and ≤80 years old；
2. Subjects with stable angina, or with unstable angina, or with subacute, old myocardial infarction, or evidence of asymptomatic ischemia；
3. Subjects with left ventricular ejection fraction ≥ 30%;
4. During the study, women of childbearing age should not become pregnant or plan to become pregnant. Therefore, it is recommended that subjects use adequate contraceptive measures until (including) the end of the follow-up period；
5. Subjects should have sufficient compliance and agree to receive follow-ups in month-1, 6, 9 and 12, and follow-up visit in year-2. It is required to perform angiography in 9 month；
6. Subjects should volunteer to participate in this study, and sign the written informed consent form, and understand all risks and benefits in the informed consent document.

   Related to the diseases:
7. The target lesion is primary, in situ coronary artery lesion, located on 1 or 2 different coronary vessels, and the number of target lesions on each coronary vessel does not exceed 1；
8. Reference vessel diameter between 2.0 mm and 2.75 mm；
9. Non-target vascular lesions need to be treated with interventional therapy first (must be treated at the same time), after successful treatment, random and target lesions will be treated;
10. Preoperative diameter stenosis must be ≥70% or ≥50% with ischemia; (visual inspection)
11. Each target lesion can only be treated with one experimental drug balloon;

Exclusion Criteria:

1. Subjects with myocardial infarction within one week, or subjects whose troponin has not returned to normal despite the onset of myocardial infarction for more than one week;
2. Subjects with severe congestive heart failure or NYHA IV heart failure;
3. Women who are pregnant or breastfeeding;
4. Subjects whose life expectancy does not exceed 1 year or who have factors that make clinical follow-up difficult;
5. Subjects with stroke within 6 months;
6. Subjects who are participating in any other clinical trials and have not reached the primary clinical endpoint;
7. Existing or history of severe liver failure, therefore not eligible for angiography;
8. Existing or history of severe renal failure (GFR<30ml/min), therefore not eligible for angiography;
9. Heart transplant;
10. Cardiogenic shock;
11. Coronary artery spasm without significant stenosis;
12. The researchers think that the subjects are not suitable for others inclusion reason;
13. Evidence of extensive thrombus in the target vessel before intervention;
14. Coronary artery bypass grafting using vein grafts;
15. Complete occlusion of the target vessel (TIMI grade 0 blood flow before operation)
16. Target vessels are distorted or have calcified lesions that cannot be pre-dilated successfully;
17. Lesions within 5 mm from the coronary artery ostia;
18. Lesions that cannot be treated with PTCA or other interventional techniques;
19. After pre-dilation of the target lesion, residual stenosis > 50% or TIMI blood flow < grade 3, and/or type C or above dissection;
20. Subjects with bleeding constitution, contraindicated anticoagulant or antiplatelet drugs;
21. Subjects who cannot tolerate aspirin and/or clopidogrel or have a history of neutropenia or thrombocytopenia, or severe liver insufficiency that prohibits clopidogrel;
22. Subjects who are known to be intolerant or allergic to heparin, contrast medium, paclitaxel, iopromide, polylactic acid-glycolic acid polymer, stainless steel, etc.;
23. Leukopenia (white blood cell count <3×109/L for more than 3 days) or neutropenia (ANC<1000 neutrophils/mm3 for more than 3 days) or history of thrombocytopenia (<100,000 platelets/mm3) subjects;
24. Subjects with a history of peptic ulcer or gastrointestinal bleeding in the past 6 months;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
In-segment diameter stenosis in target lesion(%). | 9 months
  DS% = (1 - minimum luminal diameter within the target lesion segment / reference diameter within the target lesion segment) × 100%.

SECONDARY OUTCOMES:
Technical success rate | Immediate postoperative
  defined as the successful arrival of the device to the target lesion, successful dilation, and smooth withdrawal, without the use of any additional interventional treatment methods, with residual stenosis ≤30% (estimated method), TIMI blood flow grade 3, and no grade C or higher dissection.
Lesion success rate | Immediate postoperative
  defined as residual stenosis within the target lesion segment being ≤30% (estimated method) after using any interventional treatment method, with TIMI blood flow grade 3 and no grade C or higher dissection.
Procedural success rate | during the hospitalization and no more 7 days
  defined as the absence of device-related composite endpoint events during the hospitalization period on the basis of lesion success rate
The proportion of subjects with target lesion failure. | in month-1, 6, 9, 12 ,24
  defined as the composite endpoint of cardiac death, target vessel-related myocardial infarction (TV-MI) and ischemia-driven target lesion revascularization (ID-TLR);
The proportion of subjects with patient-related composite endpoints | in month-1, 6, 9, 12 ,24
  defined as the composite endpoint of all-cause death, all myocardial infarctions, and any revascularization
Proportion of Subjects' mortality | in month-1, 6, 9, 12 ,24
Proportion of Subjects' myocardial infarction | in month-1, 6, 9, 12 ,24
Proportion of Subjects' target lesion revascularization | in month-1, 6, 9, 12 ,24
Proportion of Subjects' any coronary revascularization | in month-1, 6, 9, 12 ,24
Proportion of Subjects with Thrombotic Events as defined by ARC | in month-1, 6, 9, 12 ,24
  includes definite, probable, and unexcluded thrombus in the acute, subacute, late, and late late timeframes
Incidence Rate of All AE and SAE in subjects | in month-1, 6, 9, 12 ,24
Late Lumen Loss | 9 months
  defined as the change in minimal lumen diameter
Incidence of target lesion restenosis | 9 months
  proportion of patients with >50% diameter stenosis

CONTACTS AND LOCATIONS:
Locations (1):
- Meizhou People's Hospital (Huangtang Hospital, Meizhou Academy of Medical Sciences), Meizhou, Guangdong, China